CLINICAL TRIAL: NCT00112775
Title: A Randomized Multi-Center Open Label Study of BMS-354825 vs Imatinib Mesylate (Gleevec®) 800 mg/d in Subjects With Chronic Phase Philadelphia Chromosome-Positive Chronic Myeloid Leukemia Who Have Disease That is Resistant to Iamtinib at a Dose of 400-600 mg/d
Brief Title: BMS-354825 or Imatinib Mesylate in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia That Did Not Respond to Previous Imatinib Mesylate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000428457; UCLA-0501047-01; BMS-CA180017; EUDRACT-2004-004450-96
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2006-04

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Imatinib Mesylate

INTERVENTIONS:
Drug: dasatinib
Drug: imatinib mesylate

SUMMARY:
RATIONALE: BMS-354825 and imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This randomized phase II trial is studying BMS-354825 to see how well it works compared to imatinib mesylate in treating patients with chronic phase chronic myelogenous leukemia that did not respond to previous imatinib mesylate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 12-week major cytogenetic response (MCyR) rate in patients with imatinib mesylate-resistant Philadelphia chromosome-positive chronic phase chronic myelogenous leukemia treated with BMS-354825 vs imatinib mesylate.

Secondary

* Determine the MCyR rate prior to crossover in patients treated with these drugs.
* Determine the durability of MCyR and time to MCyR prior to crossover in patients treated with these drugs.
* Determine the complete hematologic response (CHR) rate prior to crossover in patients treated with these drugs.
* Determine the durability of CHR and time to CHR prior to crossover in patients treated with these drugs.
* Determine the major molecular response rate prior to crossover, as determined by BCR-ABL transcripts in blood during treatment using quantitative reverse transcriptase polymerase chain reaction, in patients treated with these drugs.
* Determine post-crossover efficacy endpoints in patients treated with these drugs who crossover.
* Assess health-related quality of life prior to crossover in patients treated with these drugs.
* Determine the safety and tolerability of BMS-354825 in these patients.
* Determine the pharmacokinetics of BMS-354825 in these patients.

OUTLINE: This is an open-label, multicenter, randomized, crossover study. Patients are stratified according to study site and cytogenetic response to prior imatinib mesylate (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral BMS-354825 twice daily in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression or persistent intolerance to BMS-354825 cross over to arm II after a 2-day washout period. After crossover, patients receive oral imatinib mesylate twice daily in the absence of further disease progression or unacceptable toxicity.
* Arm II: Patients receive oral imatinib mesylate twice daily in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression, intolerance to imatinib mesylate, lack of major cytogenetic response at 12 weeks, or < 30% absolute reduction in Philadelphia chromosome-positive metaphases at 12 weeks cross over to arm I after a 1-week washout period. After crossover, patients receive oral BMS-354825 twice daily in the absence of further disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at day 29, every 4 weeks for 24 weeks, every 12 weeks for the remainder of study treatment, and then at the completion of study treatment.

After the completion of study treatment, patients are followed for at least 30 days.

PROJECTED ACCRUAL: A minimum of 150 patients (100 in arm I and 50 in arm II) will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic phase chronic myelogenous leukemia (CML), meeting all of the following criteria:

  * Less than 15% blasts in peripheral blood and bone marrow
  * Less than 20% basophils in peripheral blood
  * Less than 30% blasts and promyelocytes in peripheral blood and bone marrow
  * Platelet count ≥ 100,000/mm^3 (unless thrombocytopenia is due to recent therapy)
  * No extramedullary involvement (other than liver or spleen)
* Philadelphia chromosome (Ph)-positive disease by cytogenetic analysis
* Must have developed resistant disease during prior treatment with imatinib mesylate* at a dose of 400-600 mg/day**, as defined by 1 of the following:

  * Loss of major cytogenetic response (MCyR)

    * Achieved a confirmed MCyR and subsequently no longer meets the MCyR criteria
    * Documented increase in Ph-positive metaphases by 30% on 2 cytogenetic analyses performed ≥ 4 weeks apart during treatment with imatinib mesylate
  * Loss of complete hematologic response (CHR)

    * Achieved a confirmed CHR and subsequently no longer meets the CHR criteria on all asessments over a consecutive 2-week period during treatment with imatinib mesylate
  * Continuously increasing WBC count on ≥ 2 consecutive evaluations ≥ 2 weeks apart with the final assessment showing a doubling of WBC from the nadir to ≥ 20,000/mm^3 OR an absolute increase in WBC by > 50,000/mm^3 above the lowest count after starting imatinib mesylate
  * No CHR after 3 months of treatment with imatinib mesylate at a dose of 400-600 mg/day
  * No cytogenetic response after 6 months of treatment with imatinib mesylate at a dose of 400-600 mg/day
  * No MCyR after 12 months of treatment with imatinib mesylate at a dose of 400-600 mg/day NOTE: *Imatinib mesylate does not need to be the most recent treatment for CML

NOTE: **Imatinib mesylate dose ≤ 600 mg/day

* Able to tolerate chronic administration of imatinib mesylate at the highest dose received during prior treatment

  * No imatinib mesylate-related non-hematologic toxicity ≥ grade 3
  * No grade 4 imatinib mesylate-related hematologic toxicity lasting more than 7 days
  * No imatinib mesylate-related toxicity that led to discontinuation or disruption of dosing for > 4 weeks
* No previously identified BCR-ABL mutation of 1 of the following types:

  * L248V
  * G250E
  * Q252H/R
  * Y253H/F
  * E255K/V
  * T315I/D
  * F317L
  * H369P/R
* No prior diagnosis of accelerated phase or blast crisis CML

  * Patients who previously met the criteria for accelerated phase or blast crisis CML who achieved CHR during treatment with imatinib mesylate and then subsequently progressed to chronic phase CML are not eligible
* Ineligible for or unwilling to undergo hematopoietic stem cell transplantation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* See Disease Characteristics
* No history of a significant bleeding disorder unrelated to CML, including any of the following:

  * Congenital bleeding disorder (e.g., von Willebrand's disease)
  * Acquired bleeding disorder diagnosed within the past year (e.g. acquired anti-factor VIII antibodies)

Hepatic

* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN
* Total serum or ionized calcium normal (supplementation allowed)

Cardiovascular

* Heart rate ≥ 50 beats/minute by EKG
* No myocardial infarction within the past 6 months
* No uncontrolled angina within the past 3 months
* No congestive heart failure within the past 3 months
* No diagnosed or suspected congenital long QT syndrome
* No history of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or torsades de Pointes)
* No prolonged QTc interval (i.e., > 450 msec) by EKG using Bazett's correction

  * High Bazett's correction (i.e., > 450 msec) allowed provided Fridericia correction is ≤ 450 msec
* No history of second or third degree heart block

  * Pacemaker allowed
* No uncontrolled hypertension
* No other uncontrolled or significant cardiovascular disease

Other

* Not pregnant
* No nursing during and for ≥ 3 months after study participation
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 1 month before, during, and for ≥ 3 months after study participation
* Magnesium and potassium normal (supplementation allowed)
* No serious uncontrolled medical disorder or active infection that would preclude study participation
* No dementia or altered mental status that would preclude giving informed consent
* No significant bleeding from the gastrointestinal tract within the past 6 months
* No evidence of organ dysfunction or any clinically significant deviation from normal on physical examination, vital signs, EKG, or clinical laboratory determinations unrelated to CML that would preclude study participation
* No prisoners or patients who are involuntarily incarcerated for treatment of either a psychiatric or physical (e.g., infectious disease) illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 14 days since prior interferon

Chemotherapy

* More than 14 days since prior cytarabine
* Prior or concurrent hydroxyurea for elevated WBC (i.e., WBC > 50,000/mm^3) allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 7 days since prior imatinib mesylate
* At least 7 days since prior and no concurrent low-dose aspirin (≤ 325 mg/day)
* At least 14 days since prior and no concurrent high-dose aspirin (> 325 mg/day)
* More than 14 days since prior targeted small molecule anticancer agents
* More than 28 days since prior investigational or antineoplastic agents except hydroxyurea or anagrelide
* At least 5 days or 5 half-lives (whichever is greater) since prior and no concurrent drugs that carry a risk of causing torsades de Pointes, including any of the following:

  * Quinidine
  * Procainamide
  * Disopyramide
  * Amiodarone
  * Sotalol
  * Ibutilide
  * Dofetilide
  * Erythromycin
  * Clarithromycin
  * Chlorpromazine
  * Haloperidol
  * Mesoridazine
  * Thioridazine
  * Pimozide
  * Ziprasidone
  * Cisapride
  * Bepridil
  * Droperidol
  * Methadone
  * Arsenic trioxide
  * Chloroquine
  * Domperidone
  * Halofantrine
  * Levomethadyl
  * Pentamidine
  * Sparfloxacin
  * Lidoflazine
* At least 5 days or 5 half-lives (whichever is greater) since prior and no concurrent medication that directly inhibits platelet function (except anagrelide for thrombocytosis due to CML), including any of the following:

  * Dipyridamole
  * Epoprostenol
  * Epitifibatide
  * Clopidogrel
  * Cilostazol
  * Abciximab
  * Ticlopidine
* At least 5 days or 5 half-lives (whichever is greater) since prior and no concurrent anticoagulants (e.g., warfarin, heparin, or low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, or enoxaparin])

  * Concurrent prophylactic low-dose warfarin for prevention of catheter thrombosis and heparin-flush for IV lines allowed
* No prior BMS-354825
* No concurrent CYP3A4 inhibitors or inducers, including any of the following:

  * Ketoconazole
  * Ritonavir
  * Rifampin
  * Efavirenz
* No other concurrent therapy for CML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-03

PRIMARY OUTCOMES:
Major cytogenic response (MCyR) rate at 12 weeks

SECONDARY OUTCOMES:
MCyR at any time
Duration of MCyR
Time to MCyR
Complete hematologic response rate

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Kantarjian H, Pasquini R, Levy V, Jootar S, Holowiecki J, Hamerschlak N, Hughes T, Bleickardt E, Dejardin D, Cortes J, Shah NP. Dasatinib or high-dose imatinib for chronic-phase chronic myeloid leukemia resistant to imatinib at a dose of 400 to 600 milligrams daily: two-year follow-up of a randomized phase 2 study (START-R). Cancer. 2009 Sep 15;115(18):4136-47. doi: 10.1002/cncr.24504. PMID 19536906
- [Result] Kantarjian H, Pasquini R, Hamerschlak N, Rousselot P, Holowiecki J, Jootar S, Robak T, Khoroshko N, Masszi T, Skotnicki A, Hellmann A, Zaritsky A, Golenkov A, Radich J, Hughes T, Countouriotis A, Shah N. Dasatinib or high-dose imatinib for chronic-phase chronic myeloid leukemia after failure of first-line imatinib: a randomized phase 2 trial. Blood. 2007 Jun 15;109(12):5143-50. doi: 10.1182/blood-2006-11-056028. Epub 2007 Feb 22. PMID 17317857